CLINICAL TRIAL: NCT04454541
Title: The Efficacy of Ultrasound -Guided Multifidus Cervicis Plan Block Versus Greater Occipital Nerve Block for Cervicogenic Headache
Brief Title: Efficacy of Ultrasound-Guided Multifidus Cervicis Plan Block Vs Greater Occipital Nerve Block for Cervicogenic Headache
Acronym: UBLOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abha International Private Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UBLOCK
Record Dates: First submitted 2020-05-13; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Cervicogenic Headache
Keywords: Cervicogenic Headache; Headache; Cervicis Plan Block; Occipital Nerve Block
MeSH Terms: conditions — Post-Traumatic Headache; Headache

STUDY DESIGN:
Intervention Model Description: Arm A-Greater occipital nerve block The ultrasound-guided GONB was performed to more accurately locate the nerve. The patient was asked to lie prone on the table. To locate the nerve, we searched for the occipital artery in the medial one-third of the superior nuchal line between the occipital tubercle and mastoid process.
  Arm B- Multifidus cervicus plan block group (MCPB) Patients will receive continuing low-flow non humidified nasal cannula oxygen (2 L/min) and continued intravenous infusion of Ringer's solution while respiratory signs were closely monitored during the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Greater occipital nerve block with ultrasound (Active Comparator): A-Greater occipital nerve block The ultrasound-guided GONB was performed to more accurately locate the nerve. The patient was asked to lie prone on the table. To locate the nerve, we searched for the occipital artery in the medial one-third of the superior nuchal line between the occipital tubercle and mastoid process. The scalp was cleaned with iodine. After that, the skin was sterilized, and the probe was sheathed in a sterile plastic package GONB was performed by applying the injection to the medial of the artery. A 22-gauge needle was advanced beneath the lateral border of the probe using real-time ultrasound guidance and an in-plane technique. In all patients the occipital nerve was seen medial to the artery. The injected side was determined by the patients' clinical symptoms and according to the painful side reported in their headache diaries. The patients were required to lie down for 30 minutes after the injection to avoid dizziness.
  Interventions: Procedure: Ultrasound-guided nerve block for headache management
- Multifidus cervicis plane block with ultrasound guided (Experimental): Patients placed in a lateral position with their affected side upwards. Several gel cushions were placed under their head, neck, and arm to put the neck in a stable and slightly anterior flexion position spinal level was determined by identifying the transverse process of the seventh and sixth cervical vertebrae (C7 and C6). The seventh cervical transverse process (C7) differs from the levels above by having a rudimentary anterior tubercle and a prominent posterior tubercle. After aseptic preparation of the injection area, lidocaine 1% was used to anesthetize the skin. Under continuous ultrasound guidance, the needle (22-G, 0.7 mm × 60 mm, Plexufx, B-BRAUN, Tokyo, Japan) was introduced in-plane through the skin and advanced into the fascial plane between the multifidus cervicis and semispinalis cervicis muscles for the MCP block.
  Interventions: Procedure: Ultrasound-guided nerve block for headache management

INTERVENTIONS:
Procedure: Ultrasound-guided nerve block for headache management — The study was done to compare the efficacy of two different techniques: multifidus cervicus plan block and greater occipital nerve block in treatment of refractory cervicogenic headache using ultrasound guided.

SUMMARY:
Background: Cervicogenic headache (CH) described as a chronic hemi-cranial pain resulted from a disorder of the cervical spine and its anatomic structures innervated by the C1, C2, and C3 cervical spinal nerves. Traditionally noninvasive and invasive techniques were used for treatment. Greater occipital nerve block is the most frequent peripheral nerve block invasive technique used for the management of cervicogenic headache Objectives: The study was done to compare the efficacy of two different techniques: multifidus cervicus plan block and greater occipital nerve block in treatment of refractory cervicogenic headache using ultrasound guided.

Patients and Methods: sixty patients with cervicogenic headache were recruited and diagnosed according to ICHD-ш Beta version. Divided into two group, one for greater occipital nerve block and the other for multifidus cervicis plane block with ultrasound guided.

DETAILED DESCRIPTION:
This study was done to compare the efficacy of two different techniques: multifidus cervicus plane block and greater occipital nerve block in treatment of cervicogenic headache using ultrasound guided.

This prospective study that was approved by Institutional Review Board (IRB), Mansoura Faculty of Medicine, Mansoura University, Cairo Egypt (Code Number: R/19.04.483) and all participants gave written informed consent. The procedures followed were in accordance with our protocol.

This study included patients with cervicogenic headache disorders that diagnosed according to International Classification of Headache Disorder version III (ICHD-III beta version) criteria (18)

Full clinical neurological examination was done for all patients. Blood samples for routine laboratory investigations (Complete blood count, creatinine, liver function tests, PT, APTT) were taken from all patients, electrocardiography (ECG) were done for all patients. Pain intensity was evaluated via visual analog scale (VAS) scores (0 -10). Pain intensity evaluation will be done at initial presentation then after 2 and 4 weeks, using the VAS scale for affected side of cervicogenic headache. Saturation of pulse oxygen (SpO2), all Procedures performed using ultrasound system with a 7 - 13 MHz multi-frequency transducer (LOGIQ P5; GE Healthcare).

ELIGIBILITY:
Inclusion Criteria:

History of occipital nerve injection, occipital nerve stimulation or history of surgical procedures in the occipital region,

Exclusion Criteria:

* History of allergic reaction to the substance to be applied as local anesthetic.,
* Pregnancy or lactation,
* Uncontrolled hypertension,
* Uncontrolled diabetes mellitus,
* Uncompensated congestive heart failure,
* Chronic renal failure,
* Chronic liver disease,
* Tumor and/or vascular disease,
* Inflammatory and/or infectious diseases,
* Anticoagulant or antiplatelet medication use that may interfere with the injection process were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Headache free | 30 minute post intervention

SECONDARY OUTCOMES:
Visual analog scale (VAS) | 2 Weeks
Visual analog scale (VAS) | 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zenat Eldadamony Mohamed, PhD MD, Study Chair — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Background] Dočekal, P., Keller, O., Marková, J., Opavský, J. (2006) Bolesti hlavy. In: Bolest. Rokyta, R., Kršiak, M., Kozák, J., pp. 2006; 461-477, Tigis, Praha. (in Czech). International Headache Society .The International Classification of Headache Disorders, 2nd edition. Cephalalgia. 2004; 24, 1-160 (Suppl. 1). Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. Fredriksen TA, Antonaci F, Sjaastad O. Cervicogenic headache: too important to be left un-diagnosed. J Headache Pain 2015; 16:6. Chaibi A, Russell MB. Manual therapies for cervicogenic headache: a systematic review. J Headache Pain. 2012; 13:351-359.